CLINICAL TRIAL: NCT01712100
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Irbesartan Tablets Under Fed Conditions
Brief Title: Crossover Bioequivalence Study of Irbesartan 300 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRBE-T300-PVFD-1
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- irbesartan (Experimental): 300 mg tablet
  Interventions: Drug: Irbesartan
- Avapro (Active Comparator): 300 mg tablet
  Interventions: Drug: Avapro

INTERVENTIONS:
Drug: Irbesartan
  Arms: irbesartan
Drug: Avapro
  Arms: Avapro

SUMMARY:
The objective of this study was to prove the bioequivalence of Roxane Laboratories' Irbesartan 300 mg Tablets under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 and 45 years (inclusive).
2. Voluntary consent to participate in the study.
3. Body Mass Index (BMI) between 18 and 30 (inclusive).
4. Female subjects of childbearing potential - not surgically sterile or at least 2 years postmenopausal - must agree to utilize one of the following forms of contraception from screening through completion of the study: abstinence, hormonal (oral, implant, transdermal, or injection) for at least 3 months prior to the first dose of the study, barrier (condom with spermicide, diaphragm with spermicide), IUD, or vasectomized partner (6 months minimum).
5. No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

1. A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. A history of allergic or adverse responses to Irbesartan, or any comparable or similar product.
3. Subjects who (for whatever reason) have been on an abnormal diet or have had substantial changes in eating habits within 30 days prior to study initiation.
4. Subjects must not have made a blood donation of one pint or more within 30 days prior to study initiation.
5. Subjects must not have made a plasma donation within 14 days of study initiation.
6. Participation in a clinical trial within 30 days prior to study initiation.
7. Use of any over-the-counter (OTC) medication, including vitamins, herbal products, and dietary supplements, within 7 days prior to or during the study.
8. Use of any prescription medication within 7 days prior to or during the study, with the exception of hormonal contraceptives for women of childbearing potential, or hormone replacement therapy.
9. Treatment with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, phenytoin, rifampin, rifabutin, glucocorticoids, diltiazem, ketoconazole, MAOI, antidepressants, neuroleptics, verapamil, quinidine, erythromycin, etc., within 30 days prior to or during the study.
10. Smoking or use of tobacco products within 6 months prior to or during the study.
11. Female subjects who are lactating.
12. Positive serum pregnancy test for female subjects.
13. Positive blood screen for HIV, Hepatitis B or Hepatitis C.
14. Positive screen for alcohol or drugs of abuse, and history or presence of alcoholism or drug abuse within 6 months prior to the study start.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2007-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | Blood samples will be collected in Vacutainers containing K3EDTA (1 x 7 mL) before dose and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, and 72 hours after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Jolene K Berg, MD, Principal Investigator — Worldwide Clinical Trials Drug Development Solutions (formerly CEDRA Clinical Research)
Locations (1):
- Worldwide Clinical Trials Drug Development Solutions (formerly CEDRA Clinical Research), San Antonio, Texas, United States